CLINICAL TRIAL: NCT06686446
Title: Allergic Rhinitis Improvement Through Strategic Education: The ARISE Trial
Acronym: ARISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NACE-003
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Allergy
Keywords: Allergy Rhinitis
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional, randomised trial, evaluating the impact and effectiveness of a new AR education package used in conjunction with daily INCS or INCS+INAH treatment to reduce AR-related symptomatology and improve quality of life, in comparison to the standard of care education that is currently provided. A decentralized clinical trial model will be used to facilitate and augment the recruitment of participants across different geographical locations around Australia to align with the seasonal pollen changes in various states and territories.
  Consented participants will be randomised 1:1 to either the intervention group who receive an Enhanced Education Package (EEP) which is a targeted set of patient education tools and weekly email/SMS reminders over a 6 week period, or to the control group (standard of care), which may include management by a general practitioner, specialist, pharmacist, or self-management).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Education Package (Experimental): Participants randomised to the intervention arm will receive an advanced patient education toolkit and reminders delivered by email/SMS in addition to the standard education which may include management by a general practitioner, specialist, pharmacist, or self-management.
  The EEP will contain:
  * Dosing/frequency - links for package inserts for INCS and INCS+INAH
  * Correct INCS or INCS+INAH technique - the study team will ask participants to show them the correct technique in taking their nasal spray
  * Weekly repeat reminders - these reminders will be sent via either SMS or email over a period of 6 weeks. They will instruct and remind the participant to take their INCS or INCS+INAH as per their treating clinician recommendation and why it is important to take it as instructed.
  * Education Toolkit - contains links to websites of key organisations which include educational videos and other resources
  Interventions: Behavioral: Enhanced Education Package
- Standard of care (No Intervention): Participants randomised to the control arm will receive standard of care education, which may include management by a general practitioner, specialist, pharmacist, or self-management.
  After randomisation, the study team will confirm what education the participants have received and that they can display the correct technique in taking their nasal spray. The research assistant/study nurse can re-educate the participant until the correct technique is displayed.

INTERVENTIONS:
Behavioral: Enhanced Education Package — Participants randomised to the intervention arm will receive an advanced patient education toolkit and reminders delivered by email/SMS in addition to the standard education provided by their treating clinician.
  Weekly repeat reminders - these reminders will be sent via either SMS or email over a period of 3 months. They will instruct and remind the participant to take their INCS/INAH as per their treating clinician recommendation and why it is important to take it as instructed.
  Education Toolkit - contains links to websites of key organisations including the National Allergy Council (NAC), Allergy & Anaphylaxis Australia (A&AA), Australasian Society of Clinical Immunology and Allergy (ASCIA), National Asthma Council Australia (NACA) and AusPollen which include educational videos and other resources.
  Arms: Enhanced Education Package

SUMMARY:
Allergic Rhinitis, or hay fever, is a common allergic chronic condition that affects many Australians, with its prevalence rates increasing each year due to environmental factors and affects all age groups. Evidence shows a large proportion of individuals with hay fever, whether it is seasonal, perennial (all year round) or occupational, will not seek medical help and instead rely on over the counter medications. This often leads to inadequate treatment and poor control of symptoms, impacting their quality of life, symptom burnout and economic burden.

There are effective treatments available including Intranasal Corticosteroid (INCS) sprays or combination INCS + Intranasal Antihistamine (INAH) sprays, but they need to be used correctly and as directed for best results. Previous studies have shown that many adults and children who use INCS+INAH do not know the right way to use them because they are not provided with enough education and awareness. Studies also show that adolescents and young adults are more likely to not follow their treatment plan because they worry about minor side effects INCS or INCS+INAH can cause, and misconceptions that can come from a lack of education. However, these concerns can be avoided if they are guided and educated on the correct techniques, knowledge through repeat education.

DETAILED DESCRIPTION:
This study will be a prospective decentralised interventional trial that will address the following research question: In adolescents and young adults with moderate to severe AR does six weeks of a targeted intervention package of patient education tools reduce AR symptoms and positively impact other patient reported outcomes compared to standard AR management?

Trial participants aged 14-29 will be recruited via both direct to patient advertising and participating recruitment sites (for example, allergy specialists, hospital outpatient clinics and general practitioners), located across Australia.

Participants will be currently experiencing AR symptoms of at least moderate to severe severity (as per ARIA guidelines), have a previous positive SPT and/or sIgE to at least one aeroallergen, and will be using or about to start using either a INCS or a combined INCS+INAH spray.

Patients interested in participating in the trial will be able to register their interest via an online webform and complete a few eligibility screening questions. The central study team will then undertake an informed consent process via telehealth. As part of informed consent, participants are asked to allow the study team to request access to their skin prick test and/or sIgE results. Consented participants will be randomised 1:1 to either the intervention group who receive an Enhanced Education Package (EEP) which is a targeted set of patient education tools and weekly email/SMS reminders over a 6 week period, or to the control group (standard of care), which may include management by a general practitioner, specialist, pharmacist, or self-management). All participants will be assessed at baseline and 6 weeks post-randomisation on physical symptoms (nasal and ocular symptoms) and quality of life. A validated questionnaire to assess knowledge, attitude and practice (KAP) of nasal steroid and its uses, will also be given to all participants in each group at both timepoints. All assessment measures will be repeated at 9-months post-randomisation to look at longer term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents and young adults aged 14-29 years experiencing moderate to severe AR symptoms (defined by ARIA guidelines if AR symptoms significantly affect sleep or activities of daily living, and/or if they are considered bothersome (15)) and is using or commencing INCS or combination INCS+INAH treatment.
2. A previous positive SPT and/or sIgE to at least one aeroallergen
3. Ability to understand and comply with study requirements and provide informed consent

Exclusion Criteria:

1. Current or previous treatment for AR with aeroallergen immunotherapy (patients will be specifically asked if they have ever received subcutaneous immunotherapy (SCIT) or sublingual immunotherapy (SLIT) for aeroallergens such as pollen, house dust mite, cats, dogs and horses)

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference between the two treatment arms (experimental versus standard of care) in participant nasal symptomatology: Change in total scores 6 weeks post commencement of INCS or INAH+INCS | Baseline and 6-weeks post-randomisation
  Patient reported nasal symptomatology scores completed using the validated Total Nasal Symptom Score (TNSS) questionnaire. The TNSS questionnaire is a validated questionnaire to assess nasal symptomatology and consists of 3 questions. Total scores are calculated by adding the sum of completed items. Questions are based on a 3 point Likert scale, with scores of 6 or more indicating moderate to severe allergic rhinitis.

SECONDARY OUTCOMES:
Difference between treatment arms in participant nasal symptomatology: Change in total scores 9 months post commencement of INCS or INAH+INCS | Baseline and 9-months post-randomisation
  Patient reported nasal symptomatology scores completed using the validated Total Nasal Symptom Score (TNSS) questionnaire. The TNSS questionnaire is validated questionnaire to assess nasal symptomatology and consists of 3 questions. Total scores are calculated by adding the sum of completed items. Questions are based on a 3 point Likert scale, with scores of 6 or more indicating moderate to severe allergic rhinitis.
Change between treatment arms in participant ocular symptomatology | Baseline, 6 weeks post randomisation and 9 months post randomisation
  Patient reported ocular symptomatology scores completed using the Total ocular symptom score (TOSS) questionnaire. The TOSS questionnaire is validated questionnaire to assess ocular symptomatology and consists of 3 questions. Total scores are calculated by adding the sum of completed items. Questions are based on a 3 point Likert scale, with scores of 6 or more indicating moderate to severe allergic rhinitis.
Mean change between treatment arms in Quality of Life Scores using the Rhinitis Control Assessment Test (RCAT) | Baseline, 6 weeks post randomisation, 9 months post randomisation
  The Rhinitis Control Assessment Test (RCAT) questionnaire is validated questionnaire to assess Allergy Rhinitis symptoms and impact on quality of life. It is completed by participants and consists of 6 questionnaires. Total scores are calculated by adding the sum of completed items. Questions are based on a 5 point Likert scale, with scores of 21 or less indicating greater impact on quality of life.
Change between treatment arms in participant knowledge, attitude and practice on nasal steroid and its uses | Baseline, 6 weeks post randomisation and 9 months post randomisation
  The Allergic Rhinitis Knowledge, Attitude and Practice (KAP) are disease-specific questionnaire for participants with allergy rhinitis. The KAP is completed by participants and consists of 12 items over 3 domains (knowledge, attitudes and practice). The knowledge section is based on a 3 point Likert scale using Yes, Not sure and No. Attitude section is based on a 6 point Likert scale and total and scores are calculated by the sum of completed items. Higher scores indicating positive attitudes towards their health condition. Practice section is based on a 5 point Likert scale and total and scores are calculated by the sum of completed items. Higher scores indicating excellent practice in treating their health condition. Each section will be scored separately.
Change between treatment arms in total scores for participant INCS or INCS+INAH application technique | Baseline, 6 weeks and 9 months post randomisation
  INCS/INAH application technique will be observed by the study nurses/research assistants and scored using the current Australasian Society of Clinical Immunology and Allergy (ASCIA) Guidelines checklist. There are total of 6 steps and each step achieved will be given a score of 1. If not achieved a score of 0 will be given. Total scores are calculated by the sum of all 6 steps. Higher scores indicating excellent knowledge and practice in technique.
Change between treatment arms in participant engagement with educational resources from baseline to 6 weeks | Baseline then at 2 weeks, 4 weeks, 6 weeks
  Participants randomized to the EEP will be asked about education resources at baseline and if they are currently using them. Each participant will receive education toolkit with links to the current educational resources available via eNewsletters every 2 weeks during the 6 week intervention window. Campaign monitor analytics will be used to record number of clicks on the educational resources provided. Higher the clicks indicates greater participant engagement.

OTHER OUTCOMES:
Exploratory objective: Effect of factors influencing the effectiveness of the Enhanced Education Package: A percentage total is assigned to the factors studied | Baseline and 6 weeks post randomisation
  Baseline AR severity (TNSS), type of AR (seasonal or perennial), baseline KAP, demographics (including age, rurality, ethnicity, language), sensitisation and allergy history, on TNSS will be assessed and calculated as a percentage in influencing the scores relating to the effectiveness use of the enhanced education package. Higher percentage indicates greater influence.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten M Perrett, MBBS, FRACP, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
After the data has been cleaned and database has been locked, the de-identified data and if consented, personal identifying information, will be shared to National Allergy Centre of Excellence (NACE) Allergy BioRepository via a safe and secure mechanism, for storage and use in future allergy research.
Supporting Information: CSR, Analytic Code
Time Frame: On completion of the ARISE study, de-identified data, encrypted with NACE unique identifier codes and secure linkage key tokens, will be transferred to the ALBI platform, for storage, integration and sharing for future HREC-approved allergy research purposes. Data once in ALBI remains indefinitely.
Access Criteria: ALBI will only provide researchers with non-identifiable information related to the specific project, following the Scientific Access Framework. Researchers need to apply for access to ALBI data. This is done via NACE email: nace@mcri.edu.au. Once approved, data will be made available to the researchers by logging in through a secure research platform. Researchers will not have access to the entire ALBI system as they will be provided extracts from ALBI of non-identifiable information related to their specific project upon request and approvals. Information will only be shared with ethically approved future allergy research studies. For more information about the data deidentification process.
URL: https://www.nace.org.au/

REFERENCES:
- See also: ARISE trial information — https://www.nace.org.au/research/respiratory-allergy/